CLINICAL TRIAL: NCT05187442
Title: The Experiences of Erotic and Sexual Risk of Transgender Men: Exploratory Research Design
Status: Completed | Type: Observational
Sponsor: National Taiwan University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Piao-Yi Chiou, Associate Professor, National Taiwan University
Other Study IDs: 20210HS3001
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Transgender Persons; Sexual Health
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire, interview — The first stage is an online questionnaire survey. A total of 321 TMs were recruited. The time of online questionnaire is about 10-15 minutes to get a preliminary understanding of the erotic and sexual risk experience of TM in Taiwan. In the second stage, focus groups and in-depth interviews will be conducted, 2 hours of each group and interview. A total of 29 transgender man and women, and non-binary participants were recruited.

SUMMARY:
Transgender male (TM) is the minority and difficult to reach-up group. Therefore, there is a lack of research on private issues involving TM, such as sex, eroticism, and sexual risk behavior. This study focuses on TM as the research participant, based on Milton Mayeroff's caring theory, to understand the TM's erotic culture and the sexual risks behavior, to evaluate the need for subsequent sexual health care. The research method is a mixed methods research of explanatory design, which recruits participants through purposive sampling and respondent-driven sample (RDS) methods. The first stage is an online questionnaire survey. A total of 321 TMs were recruited. The time of online questionnaire is about 10-15 minutes to get a preliminary understanding of the erotic and sexual risk experience of TM in Taiwan. In the second stage, focus groups and in-depth interviews will be conducted, 2 hours of each group and interview. A total of 29 transgender man and women, and non-binary participants were recruited. The recruitment will be stop when the data are saturated. The analysis of both quantitative and qualitative data can get an in-depth understanding of sex, eroticism, and sexual risk, and violence experiences of the participants. The research results are important for improving the awareness and identification of sexual risk and the assessment of sexual health care needs of TM in health care profession. The results also serve as a reference guide for the development of care needs on sexual health care and anti-violence of transgender people, and for the implement of a gender-friendly environment for medical care.

ELIGIBILITY:
First stage:

Inclusion Criteria:

1. People who used to or currently self-identified as transgender men, regardless of whether they have sex reassignment surgery.
2. Be over 20 years old.
3. Citizen and live in Taiwan.

Exclusion Criteria:

1. Not self-identify as transgender men
2. Younger than 20 years old
3. Not citizen and not live in Taiwan.

Second stage

1. People who used to or currently self-identified as transgender men, transgender woman or non-binary, regardless of whether they have gender-affirming surgery.
2. Be over 20 years old.
3. Citizen and live in Taiwan.

Exclusion Criteria:

1. Not self-identify as transgender men, transgender woman or non-binary.
2. Younger than 20 years old
3. Not citizen and not live in Taiwan.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender:transgender men
Study Population: 1. The personal network of the research team is used to search for eligible TMs via social media platforms, such as Facebook (FB), Instagram (IG), and group of Line app.
  2. The recruitment materials will be published on transgender communities, social media platforms, non-governmental organizations, and YouTube, etc., to recruit the participants.
  3. The participants who finished the online questionnaire will be encourage to invite and transfer their network who meet the inclusion criteria via Line app or email address to our research team.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing of National Taiwan University, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: TM participants were recruited using Respondent-Driven Sampling (RDS), starting with individuals who expressed willingness to participate. These participants then referred others to ensure heterogeneity and diversity in the sample. In Stage 2, qualitative interviews with Tran woman and non-binary individuals were conducted using snowball and purposive sampling methods. These groups served as experiential references to complement the qualitative and survey findings from the TM group.
Groups:
- Transgender: Transgender individuals
Period: Stage 1: Online Survey
Arm/Group | Transgender
Started | 321
Completed | 321
Not Completed | 0
Period: Stage 2: Focus Groups
Arm/Group | Transgender
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Transgender individuals. The "Age" data were not collected for participants in Stage 2.
Groups:
- Stage 1: Online Survey Transgender; Stage 2: Focus Groups Transgender: Transgender individuals
- Total: Total of all reporting groups
Arm/Group | Stage 1: Online Survey Transgender | Stage 2: Focus Groups Transgender | Total
Number analyzed (Participants) | 321 | 29 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] — The "Age" data were not collected for participants in Stage 2. Population: The "Age" data were not collected for participants in Stage 2.
  years
    number analyzed (Participants) | 321 | 0 | 321
    (all) | 29.81 (5.764) |  | 29.81 (5.764)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 269 | 9 | 278
  Non-binary | 32 | 10 | 42
  Other | 20 | 0 | 20
  Trans woman | 0 | 10 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 321 | 29 | 350
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 321 | 29 | 350

OUTCOME MEASURES:

1. Primary Outcome: Experience of Erotic and Sexual Risk of Transgender Men(Demographic Data, Transgender Affirmation Questionnaire)
Description: After signing the online consent form, fill out the demographic information form and transgender affirmation questionnaire on Google Forms to calculate population proportions and averages.(First stage)
Time Frame: At time of entry into study
Population: Transgender individuals
Measure: Count of Participants; unit: Participants
Arm/Group | Transgender
Number analyzed (Participants) | 321
Participants
  Gender identity :male | 269
  Gender identity:other | 52
  Sexual orientation:heterosexual | 166
  Sexual orientation:gay | 37
  Sexual orientation:bisexuality | 77
  Sexual orientation:pansexuality | 33
  Sexual orientation:asexuality | 6
  Sexual orientation:other | 2
  Transgender Status:gender dysphoria | 164
  Transgender Status:GAHT | 169
  Transgender Status: chest reconstruction surgery | 138
  Transgender Status: GAS | 43
  Transgender Status: genital reconstruction | 6

2. Primary Outcome: Ages of Transgender Men
Description: After signing the online consent form, fill out the ages on Google Forms to calculate population proportions and averages.(First stage)
Time Frame: At time of entry into study
Measure: Mean (Full Range); unit: years
Arm/Group | Transgender
Number analyzed (Participants) | 321
years | 29.81 [20 to 47]

3. Primary Outcome: Experience of Erotic and Sexual Risk of Transgender Men (Short Sexual Well Being Scale)
Description: After signing the online consent form, fill out the Short Sexual Well Being Scale on Google Forms to calculate population proportions and averages.(First stage)
  Short Sexual Well Being Scale:There are a total of five questions, using a Likert 7 lit table, with scores ranging from 5 (minimum) to 35 (maximum), with the higher the score, the better Sexual Well Being.
  1. I disagree completely, 2. I disagree, 3. I disagree a little, 4. Neutral, 5. I somewhat agree, 6. I agree, 7. I completely agree
Time Frame: At time of entry into study
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Transgender
Number analyzed (Participants) | 321
score on a scale | 20.42 [5 to 30]

4. Primary Outcome: Experience of Erotic and Sexual Risk of Transgender Men (STIs Prevention Questionnaire)
Description: After signing the online consent form, fill out the STIs prevention questionnaire on Google Forms to calculate population proportions and averages.(First stage)
Time Frame: At time of entry into study
Measure: Count of Participants; unit: Participants
Arm/Group | Transgender
Number analyzed (Participants) | 321
Participants
  HIV screening | 69
  HPV screening | 43
  Pap smear | 55
  STIs | 46
  used PrEP within a year | 3

5. Primary Outcome: Violence Experience of Transgender (Experiences of Abuse & Coping Strategies)
Description: In the second stage, focus groups and in-depth interviews will be conducted, 2 hours of each group and interview.
  The interview outline was revised based on the questionnaire analysis results, and TMs who met the research requirements were selected from the questionnaire respondents to conduct physical focus groups or in-depth face-to-face or video semi-structured interviews on the theme of violence experience. We also recruited Trans woman and non-binary gender groups to conduct focus groups and in-depth interviews to compare the differences in their experiences of violence.
  The data were categorized into two main themes:Experiences of Abuse & Coping Strategies.
Time Frame: months3-6(In the second stage)
Measure: Count of Participants; unit: Participants
Arm/Group | Transgender
Number analyzed (Participants) | 29
Participants
  Experiences of Abuse:verbal abuse | 20
  Experiences of Abuse:physical violence | 6
  Experiences of Abuse:sexual violence | 18
  Experiences of Abuse:microaggression | 19
  Experiences of Abuse:Forced to come out | 8
  Coping Strategies:avoiding crowds | 26
  Coping Strategies:compromise requirements | 11
  Coping Strategies:fits the stereotype | 6
  Coping Strategies:communication explanation | 9
  Coping Strategies:advance explanation | 11
  Coping Strategies:initiative | 6
  Coping Strategies:change mindset | 19
  Coping Strategies:social welfare and psychological assistance | 11
  Coping Strategies:legal assistance | 4
  Coping Strategies:peer support | 9

ADVERSE EVENTS:
Time Frame: Quantitative Research: From the point when research participants signed the informed consent and completed the questionnaire to the distribution of vouchers, we tracked participants for approximately one year, with no adverse events reported. Qualitative Research: From the point when research participants signed the informed consent and participated in focus groups to the distribution of vouchers, we tracked participants for approximately 6 months, with no adverse events reported.
Description: Due to the cross-sectional non-interventional nature of Stage 1, participants will not be at risk for Serious Adverse Events, at risk for All-Cause Mortality, and at risk for Other (Not Including Serious) Adverse Events.
  Stage 2 underwent manual evaluation and follow-up, and no adverse events were reported.
Arm/Group | Transgender
All-Cause Mortality (participants affected / at risk) | 0/350
Serious Adverse Events (participants affected / at risk) | 0/350
Other Adverse Events (participants affected / at risk) | 0/350

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT05187442/Prot_SAP_000.pdf